CLINICAL TRIAL: NCT05747924
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Exploratory Efficacy of AOC 1020 Administered Intravenously to Participants With Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Phase 1/2 Study of AOC 1020 in Participants With Facioscapulohumeral Muscular Dystrophy (FSHD)
Acronym: FORTITUDE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOC 1020-CS1
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: FSHD; FSHD1; FSHD2; FMD; FMD2; Fascioscapulohumeral Muscular Dystrophy; Fascioscapulohumeral Muscular Dystrophy Type 1; Fascioscapulohumeral Muscular Dystrophy Type 2; Dystrophies, Facioscapulohumeral Muscular; Dystrophy, Facioscapulohumeral Muscular; Facioscapulohumeral Muscular Dystrophy 1; Facioscapulohumeral Muscular Dystrophy 2; Facio-Scapulo-Humeral Dystrophy; Atrophy, Facioscapulohumeral; Atrophies, Facioscapulohumeral; Facioscapulohumeral Atrophy; Muscular Dystrophies; Muscular Dystrophy, Facioscapulohumeral; FSH Muscular Dystrophy; Landouzy Dejerine Dystrophy; Landouzy-Dejerine Muscular Dystrophy; Dystrophies, Landouzy-Dejerine; Dystrophy, Landouzy-Dejerine; Landouzy-Dejerine Syndrome; Muscular Dystrophy, Landouzy Dejerine; Progressive Muscular Dystrophy; FSH
Keywords: FORTITUDE; Avidity; Avidity Biosciences; AOC 1020
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Facioscapulohumeral Muscular Dystrophy 1B; Muscular Dystrophies; Facioscapulohumeral muscular dystrophy 1a | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AOC 1020 Regimen 1 (Experimental): Cohort A: AOC 1020 Dose Regimen 1; Five doses administered intravenously over 9 months
  Interventions: Drug: AOC 1020
- AOC 1020 Regimen 2 (Experimental): Cohort B1: AOC 1020 Dose Regimen 2; Five doses administered intravenously over 9 months
  Interventions: Drug: AOC 1020
- AOC 1020 Regimen 3 (Experimental): Cohort C: AOC 1020 Dose Regimen 3; Eight doses administered intravenously over approximately 10 months
  Interventions: Drug: AOC 1020
- Placebo (Saline) Regimen 1 (Placebo Comparator): Cohort A & B: Placebo; Five doses administered intravenously over 9 months
  Interventions: Drug: Placebo
- Placebo (Saline) Regimen 2 (Placebo Comparator): Cohort C: Placebo; Eight doses administered intravenously over approximately 10 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOC 1020 — AOC 1020 will be administered via intravenous (IV) infusion
  Arms: AOC 1020 Regimen 1; AOC 1020 Regimen 2; AOC 1020 Regimen 3
Drug: Placebo — Placebo will be administered via intravenous (IV) infusion
  Other Names: Saline
  Arms: Placebo (Saline) Regimen 1; Placebo (Saline) Regimen 2

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Exploratory Efficacy of AOC 1020 Administered Intravenously to Participants with Facioscapulohumeral Muscular Dystrophy (FSHD)

DETAILED DESCRIPTION:
AOC 1020-CS1 is a first-in-human, 3-part, multi-center, Phase 1/2, randomized, double-blind, placebo-controlled study designed to evaluate safety, tolerability, pharmacokinetics and to explore pharmacodynamics and efficacy of single and multiple-doses of AOC 1020 administered intravenously in participants with FSHD Type 1 (FSHD1) and FSHD Type 2 (FSHD2).

Cohort A comprises a placebo-controlled dose titration cohort (Cohort A1) which includes a nested single and multiple dose schedule. Cohort B comprises a placebo-controlled, nested single ascending dose (SAD)/multiple ascending dose (MAD) cohort (Cohort B1). Cohort C comprises a randomized, placebo-controlled, expansion cohort (Cohort C1). For each of Cohorts A, B, and C the study duration is 12 months as the active treatment period is approximately 9 months for Cohorts A & B and approximately 10 months for Cohort C followed by a 12-week follow-up period for Cohorts A & B and a 7-week follow-up period for Cohort C. Once participants have completed active treatment with follow-up through 12 months, they may have the option to participate in a planned open-label extension. If patients do not enroll in the open-label extension, they will be followed for 12-weeks after their last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* FSHD1 or FSHD2 diagnosis confirmed by documented genetic testing (testing provided by Sponsor)
* Ambulatory and able to walk 10 meters (with or without assistive devices such as one cane, walking stick or braces)
* At least 1 muscle region suitable for biopsy (testing provided by Sponsor)
* Muscle weakness in both upper and lower body, as determined by Investigator

Exclusion Criteria:

* Pregnant or intends to become pregnant while on study, or active breastfeeding
* Unwilling or unable to continue to comply with contraceptive requirements
* Body mass index (BMI) >35.0 kg/m2 at Screening
* History of muscle biopsy within 30 days of the screening biopsy or planning to undergo any nonstudy muscle biopsies over the duration of the study
* History of bleeding disorders, significant keloid, or other skin or muscle conditions (e.g., severe muscle wasting) that, in the opinion of the Investigator, makes the participant unsuitable for serial muscle biopsy
* Anticipated survival less than 2 years
* Blood or plasma donation within 16 weeks of Study Day 1
* Any contraindication to MRI
* Any abnormal lab values, conditions or diseases that, in the opinion of the investigator or Sponsor, would make the participant unsuitable for the study or could interfere with participation or completion of the study
* Treatment with any investigative medication within 1 month (or 5 half-lives of the drug, whichever is longer) of Screening

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Cohorts A & B) | Through study completion, up to Day 365
Change in DUX4-regulated gene expression in muscle biopsies (Cohort C) | Day 120
Change in a circulating biomarker of FSHD disease biology (Cohort C) | Day 120

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters of AOC 1020 (Cohorts A & B) | Through study completion; up to Day 365
  Observed maximum concentration
Plasma pharmacokinetic (PK) parameters of AOC 1020 (Cohorts A & B) | Through study completion; up to Day 365
  Observed half-life
Plasma pharmacokinetic (PK) parameters of AOC 1020 (Cohorts A & B) | Through study completion; up to Day 365
  Observed area under the curve
Muscle drug concentration (Cohorts A, B & C) | Day 120
  Concentration of siRNA component in skeletal muscle
Change in DUX4-regulated gene expression in muscle biopsies (Cohort C) | Day 120
% Change in circulating creatine kinase (Cohort C) | Through study completion; up to Day 365

CONTACTS AND LOCATIONS:
Locations (17):
- United States (14):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- University of Ottawa, Ottawa, Ontario, Canada
- United Kingdom (2):
  - University College London, London
  - University of Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Avidity Biosciences Website — https://www.aviditybiosciences.com/
- See also: FORTITUDE Study Website — https://fortitude-study.com/